CLINICAL TRIAL: NCT05239910
Title: An Open Label, Phase II Study to Evaluate the Efficacy and Safety of Tenalisib (RP6530), Given With Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) Therapy for Front Line Treatment in Patients With Peripheral T-cell Lymphoma
Brief Title: Study to Evaluate the Efficacy and Safety of Tenalisib, Given With CHOP Therapy for Front Line Treatment in Patients With PTCL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in development plan
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP6530+CHOP-2103
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Tenalisib; RP6530; PI3K
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenalisib 400 mg BID and CHOP (Experimental)
  Interventions: Drug: Tenalisib
- Tenalisib 800 mg BID and CHOP (Experimental)
  Interventions: Drug: Tenalisib

INTERVENTIONS:
Drug: Tenalisib — Tenalisib will be administered orally twice daily in a 21-day cycle for 26 cycles (from cycle 1 to cycle 26), CHOP will be administered for 6 cycles (from Cycle 4 to Cycle 9) on Days 1 to 5 of each cycle.

SUMMARY:
This is a phase II open label, two-arm parallel design study of T-CHOP in patients with treatment naïve PTCL. Two doses of tenalisib (400 mg BID and 800 mg BID) will be evaluated in separate groups (Group 1: 400 mg BID and Group 2: 800mg BID) when given with standard regimen of CHOP, followed by single agent maintenance treatment with tenalisib for 1 year. Recruitment of 20 patients each will be done in both groups in parallel.

All eligible patients will start with a run-in period, in which single agent tenalisib will be administered for 3 cycles of 21 days each. Post run-in period, all patients will proceed to receive tenalisib and CHOP regimen for next 6 cycles. After completion of 6 cycles of T-CHOP treatment, maintenance therapy with tenalisib will be initiated in patients showing CR and PR. These patients will continue to receive single agent tenalisib for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of full informed consent prior to any study-specific procedures.
2. Pathologically confirmed diagnosis of PTCL according to WHO 2016 classification criteria EXCEPT following subtypes:

   * ALK-positive anaplastic T-cell lymphoma; CD30+ PTCL (who are eligible for BV and CHOP combination); extra-nodal NK/T-cell lymphoma, nasal type; HTLV1- associated lymphoma; primary cutaneous anaplastic T-cell lymphoma, T-cell lymphoma with only skin involvement
3. Disease status is defined as treatment naïve patients with PTCL who have not received prior systemic therapy for lymphoma.
4. Must have ECOG performance status ≤ 2
5. Patients must have measurable disease defined as at least one bi-dimensional measurable lesion assessed radiologically with a minimum measurement of > 1.5 cm in the longest diameter.
6. Patients must be fit to receive full-dose CHOP Therapy.
7. Adequate bone marrow, liver and renal functions

Exclusion Criteria:

1. Patients who have received prior systemic therapy for lymphoma or are receiving anticancer therapy including any investigational therapy (e.g., chemotherapy, biologic therapy, hormonal therapy).
2. Patients with known Central Nervous System (CNS) lymphoma or CNS involvement by lymphoma.
3. Active uncontrolled systemic fungal, bacterial or viral infection
4. Patient with ongoing or significant cardiac disease in last 6 months which according to the investigator can impact study participation
5. Patients with co-morbidities/complications
6. Known history of severe liver injury/disease
7. Active viral infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. and history of severe cutaneous reactions
8. Patient with any other active malignancy at the time of screening except for adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin,
9. Hypersensitivity to the active substance or to any of the excipients.
10. Pregnancy or lactation.
11. Concurrent medications or substance, the example of these treatment includes strong inhibitors or inducer of CYP3A4 enzyme or substrate of CYP3A4 with narrow therapeutic index.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate at the end of T-CHOP treatment. | 9 months
  CR rate is defined as the percentage of patients showing complete response as assessed by the Investigator according to the Lugano Classification.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) at the end of T-CHOP treatment. | 9 months
  ORR is defined as sum of CR and PR rates, as assessed by the Investigator according to the Lugano Classification
Duration of Response (DoR), | 3 years
  The duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Progression-Free Survival (PFS) | 3 years
  PFS is defined as the duration of time from start of treatment to time of documentation of progression or death from any cause
Overall Survival (OS) | 3 years
  OS is defined as the duration of time from start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No